CLINICAL TRIAL: NCT01145417
Title: An Open-Label, Extension Safety Trial Of Pregabalin In Subjects With Neuropathic Pain Associated With HIV Neuropathy (Pregabalin A0081251)
Brief Title: Pregabalin Trial In HIV Neuropathic Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081251
Record Dates: First submitted 2010-06-07; First posted 2010-06-16 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2013-05

CONDITIONS: HIV-1 Infection; Neuropathic Pain
Keywords: peripheral neuropathic pain; pregabalin; safety
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Lyrica) (Experimental)
  Interventions: Drug: pregabalin (Lyrica)

INTERVENTIONS:
Drug: pregabalin (Lyrica) — 150 mg-600 mg/day (twice daily)

SUMMARY:
This study examines the safety of pregabalin over a 6 month period in patients with neuropathic pain associated with HIV infection as an extension of another trial that tests the efficacy of pregabalin.

DETAILED DESCRIPTION:
The parent double blind study was stopped at interim analysis due to lack of efficacy and therefore this open label extension study was also terminated simultaneously on April 2, 2012; the termination was unrelated to any safety findings that could impact patient health.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the preceding A0081244 double-blind trial and completed at least through Visit 9 of that trial.

Subjects with painful distal sensory polyneuropathy (DSP) interested in treatment based on investigator's clinical judgment.

Subjects who had acceptable tolerability of study drug in A0081244.

Exclusion Criteria:

* Clinically significant or unstable conditions that, in the opinion of the investigator, would compromise participation in the study. This includes, for example, medical conditions such as, but not limited to: hepatic, renal, respiratory, hematological, immunological, cardiovascular diseases, arrhythmia, inflammatory or rheumatologic disease, active infections, symptomatic peripheral vascular disease, psychiatric illness, and untreated endocrine disorders.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Active Acquired Immune Deficiency Syndrome (AIDS)- defining Opportunistic Infection (OI) that requires hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (10):
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Providence Clinical Research, Burbank, California
  - Desert Medical Group, Inc., dba Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Desert Medical Group, Inc., dba Desert Oasis Helathcare Medical Group, Palm Springs, California
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - Neuroscience Consultants, LLC, Aventura, Florida
  - South Florida Medical Research, Aventura, Florida
  - Mount Sinai School of Medicine, New York, New York
- Colombia (2):
  - Riesgo de Fractura S.A., Bogota D.C., Cundinamarca
  - Asistencia Cientifica de Alta Complejidad, Bogota, Cundinamarca
- India (3):
  - Surakshaka Multispeciality Hospital, Hyderabad, Andhra Pradesh
  - Infectious Disease Clinic, Ahemdabad, Gujarat
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
- Hospital Nacional Dos de Mayo, Lima, Peru
- RCMI-Clinical Research Center, Rio Piedras, Puerto Rico
- South Africa (10):
  - MediSynergy, Port Elizabeth, Eastern Cape
  - Worthwhile Clinical Trials (WWCT), Lake View Hospital, Benoni, Gauteng
  - Toga Laboratory, Johannesburg, Gauteng
  - Drs Essack and Mitha, Johannesburg, Gauteng
  - Pretoria West Hospital, Pretoria West, Gauteng
  - Dr J. Reddy's Surgery, KwaDukuza, KwaZulu-Natal
  - University of Cape Town, Cape Town, Western Cape
  - Synapta Clinical Research Centre, Durban
  - Paarl Research Center, Paarl
  - Be Part Yoluntu Centre, Paarl
- Thailand (2):
  - South East Asia Research Collaboration with Hawaii, Bangkok
  - Neurology unit, Department of Medicine,, Bangkok

REFERENCES:
- [Derived] Simpson DM, Rice AS, Emir B, Landen J, Semel D, Chew ML, Sporn J. A randomized, double-blind, placebo-controlled trial and open-label extension study to evaluate the efficacy and safety of pregabalin in the treatment of neuropathic pain associated with human immunodeficiency virus neuropathy. Pain. 2014 Oct;155(10):1943-54. doi: 10.1016/j.pain.2014.05.027. Epub 2014 Jun 4. PMID 24907403
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081251&StudyName=Pregabalin%20Trial%20In%20HIV%20Neuropathic%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following completion of Visit 9 (Day 57) of double-blind trial A0081244 (NCT01049217), participants who met eligibility criteria initiated open-label treatment in the current trial A0081251 (NCT01145417).
Groups:
- Pregabalin-Pregabalin: Participants who received pregabalin during double-blind trial A0081244 (NCT01049217), received pregabalin capsule at a starting dose of 75 milligram (mg) orally twice daily, dose adjusted for optimizing pain control based on investigators discretion to allow maximum total dose of 300 mg twice daily for 6 months. Participants underwent an end-of-study medication taper over a 1-week period.
- Placebo-Pregabalin: Participants who received placebo matched to pregabalin during double-blind trial A0081244 (NCT01049217), received pregabalin capsule at a starting dose of 75 mg orally twice daily, dose adjusted for optimizing pain control based on investigators discretion to allow maximum total dose of 300 mg twice daily for 6 months. Participants underwent an end-of-study medication taper over a 1-week period.
Period: Overall Study
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Started | 108 | 109
Completed | 67 | 62
Not Completed | 41 | 47
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by sponsor | 35 | 43
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin | Total
Number analyzed (Participants) | 108 | 109 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (8.8) | 43.5 (7.9) | 42.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 68 | 139
  Male | 37 | 41 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent (TE) Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after last dose of study treatment
Population: Safety population (SAF) included all participants who signed the informed consent, had exposure to open label study drug and had at least one safety assessment.
Measure: Number; unit: participants
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 108 | 109
participants
  AEs | 67 | 70
  SAEs | 4 | 3

2. Secondary Outcome: Number of Participants Who Were Employed or Unemployed Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which SHP affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a Human Immunodeficiency Virus (HIV) neuropathy pain. Number of participants who responded "Yes/No" to Question 1: Are you currently employed (working for pay)? are reported.
Time Frame: Baseline, Week 24
Population: Intent to Treat (ITT) population: all enrolled participants who had at least one dose of open label study drug. 'N' (number of participants analyzed) signifies participants evaluable for this measure. Here 'n' signifies participants evaluable at given time point for each arm group, respectively.
Measure: Number; unit: participants
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 103 | 104
participants
  Baseline, employed (n=52,51) | 12 | 11
  Baseline, unemployed (n=52,51) | 40 | 40
  Week 24, employed (n=103,104) | 35 | 27
  Week 24, unemployed (n=103,104) | 68 | 77

3. Secondary Outcome: Absenteeism and Presenteeism Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which SHP affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a HIV neuropathy pain. Question 2 and 3 assesses absenteeism as: Hours of work missed in past 7 days due to leg/foot pain or other reason, respectively. Question 4 assesses presenteeism as: Hours of work performed in past 7 days.
Time Frame: Baseline, Week 24
Population: ITT population: all enrolled participants who had at least one dose of open label study drug. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here 'n' signifies participants evaluable at given time point for specific question for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 35 | 28
hours
  Baseline, hours missed,leg/foot pain (n=12,11) | 2.25 (6.877) | 0.82 (2.401)
  Baseline, hours missed,other reason (n=12,11) | 3.42 (6.501) | 0.91 (1.700)
  Baseline, hours worked (n=12,11) | 35.58 (15.163) | 30.36 (18.112)
  Week 24, hours missed,leg/foot pain (n=35,28) | 2.17 (4.956) | 2.32 (8.533)
  Week 24, hours missed,other reason (n=35,28) | 9.20 (21.604) | 7.71 (14.976)
  Week 24, hours worked (n=35,28) | 41.51 (20.034) | 34.86 (21.329)

4. Secondary Outcome: Productivity and Activity Impairment Assessed by Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) Questionnaire
Description: WPAI: 6-question participant rated questionnaire to determine the degree to which SHP affected work productivity while at work and affected activities outside of work. It assesses amount of absenteeism, presenteeism and daily activity impairment attributable to a HIV neuropathy pain. Question 5 and 6 assesses: How much leg/foot pain affect productivity and daily activity, respectively in past 7 days? on 11-point scale, where 0 (not affected/no impairment) to 10 (completely affected/impaired).
Time Frame: Baseline, Week 24
Population: ITT population: all enrolled participants who had at least one dose of open label study drug. 'N' (number of participants analyzed) signifies participants evaluable for this measure. Here 'n' signifies participants evaluable at given time point for specific question for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 103 | 104
Units on a scale
  Baseline, productivity affected (n=12,10) | 4.42 (2.843) | 2.40 (2.716)
  Baseline, daily activity affected (n=52,51) | 3.48 (2.846) | 3.47 (2.935)
  Week 24, productivity affected (n=35,29) | 2.17 (1.917) | 2.24 (2.415)
  Week 24, daily activity affected (n=103,104) | 2.51 (2.330) | 2.72 (2.653)

5. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36)
Description: SF-36 is a standardized survey evaluating 8 domains of functional health and well being: physical and social (So) functioning (Fn), physical and emotional role (role-physical [R-P], role-emotional [R-E]) limitations, bodily pain (BP), general health (GH), vitality (Vit), mental health (MnH). Two summary scores include Physical Component (Ph C) and Mental Component (Mn C). The score for a section is an average of the individual question scores. Score range for domain scores and summary scores: 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants who took at least one dose of open label study drug. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here 'n' signifies participants evaluable at given time point for specific parameter for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 103 | 104
Units on a scale
  Baseline: Ph Fn (n=51,53) | 73.14 (22.671) | 75.47 (22.729)
  Baseline: R-P (n=51,53) | 75.49 (22.873) | 71.93 (27.616)
  Baseline: BP (n=51,53) | 68.86 (20.430) | 68.87 (26.010)
  Baseline: GH (n=51,53) | 72.25 (20.369) | 68.79 (20.411)
  Baseline: Ph C (n=51,53) | 47.68 (7.268) | 46.85 (9.578)
  Baseline: Vit (n=51,53) | 71.57 (19.418) | 73.11 (17.660)
  Baseline: So Fn (n=51,53) | 78.92 (18.113) | 82.08 (18.911)
  Baseline: R-E (n=51,53) | 81.05 (20.075) | 79.87 (23.367)
  Baseline: MnH (n=51,53) | 76.27 (18.079) | 80.00 (15.411)
  Baseline: Mn C (n=51,53) | 51.41 (8.915) | 52.71 (7.763)
  Week 24: Ph Fn (n=103,104) | 70.34 (27.594) | 75.24 (25.086)
  Week 24: R-P (n=103,104) | 71.18 (24.927) | 72.96 (26.680)
  Week 24: BP (n=102,104) | 69.57 (22.550) | 72.19 (23.033)
  Week 24: GH (n=103,104) | 73.14 (19.933) | 71.31 (19.879)
  Week 24: Ph C (n=102,104) | 47.28 (8.770) | 48.48 (8.634)
  Week 24: Vit (n=103,104) | 68.51 (18.502) | 66.29 (20.039)
  Week 24: So Fn (n=103,104) | 79.98 (20.883) | 81.85 (20.304)
  Week 24: R-E (n=103,104) | 74.19 (27.029) | 75.80 (25.640)
  Week 24: MnH (n=103,104) | 76.21 (18.196) | 75.77 (18.588)
  Week 24: Mn C (n=102,104) | 50.15 (10.394) | 49.72 (9.884)

6. Secondary Outcome: Visual Analogue Scale for Pain (VAS-pain)
Description: Participants rated the severity of HIV neuropathy pain on a 0 to 100 millimeter (mm) Visual Analog Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, Week 4, 8, 12, 16, 20, 24
Population: ITT population: all enrolled participants who had at least one dose of open label study drug. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here 'n' signifies participants who were evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 107 | 108
millimeter (mm)
  Baseline (n=107,108) | 40.6 (26.55) | 40.7 (26.57)
  Week 4 (n=106,106) | 33.1 (25.14) | 33.1 (27.11)
  Week 8 (n=100,101) | 27.4 (21.01) | 27.8 (24.25)
  Week 12 (n=89,88) | 24.1 (22.41) | 23.8 (23.45)
  Week 16 (n=85,81) | 22.6 (20.82) | 22.6 (25.32)
  Week 20 (n=72,67) | 17.2 (19.18) | 17.7 (22.78)
  Week 24 (n=103,104) | 22.2 (22.54) | 23.7 (23.94)

7. Secondary Outcome: Number of Participants With Categorical Scores on Patient Global Impression of Change (PGI-C)
Description: PGI-C: participant rated instrument to measure participant's change in overall status since the start of the study, on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Number of participants in each category are reported.
Time Frame: Week 24
Population: ITT population: all enrolled participants who had at least one dose of open label study drug. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 103 | 104
participants
  Very Much Improved | 41 | 37
  Much Improved | 43 | 47
  Minimally Improved | 16 | 16
  No Change | 2 | 3
  Minimally Worse | 1 | 0
  Much Worse | 0 | 1
  Very Much Worse | 0 | 0

8. Secondary Outcome: Number of Participants With Response to Sheehan-Suicidality Tracking Scale (S-STS) Mapped to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories
Description: S-STS:8-item clinician/participant administered prospective rating scale to assess TE suicidal(Su) ideation(ID),behavior(BHV).Items 1a,2-6,7a,8 scored on 5-point Likert scale 0(not at all) to 4(extremely). Items 1,1b,7 require yes/no response. S-STS total score range 0-30. Lower score=reduced Su tendency. Responses on S-STS were mapped to Columbia Classification Algorithm of Suicide Assessment(C-CASA) as 1:Completed Su; 2: Su attempt; 3: Preparatory acts; 4: Su ID; 5: Self-injurious (SI) BHV, intent unknown; 6: Not enough information; 7: SI BHV, no Su intent; 8: Other, no deliberate self harm.
Time Frame: Baseline up to Week 25
Population: SAF included all participants who signed the informed consent, had exposure to open label study drug and had at least one safety assessment.
Measure: Number; unit: participants
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 108 | 109
participants
  Suicide attempt: 2 | 0 | 1
  Preparatory acts toward suicidal behavior: 3 | 0 | 1
  Suicidal ideation: 4 | 4 | 9

9. Secondary Outcome: Number of Participants With Response to Patient Health Questionnaire-8 (PHQ-8)
Description: PHQ-8: 8-item self-administered validated subset of PHQ-9, which comprises first 8 items of measure. Participant rated "Over past 2 weeks, how often bothered by any of following problems?": little interest in doing things(1); feeling down(2); trouble falling or staying asleep/sleeping too much(3); feeling tired(4); poor appetite/overeating(5); feeling bad about self(6); trouble concentrating(7); moving or speaking slowly or being so fidgety/moving around more than usual(8). Each item scored on scale of 0(not at all)-3(nearly every day). Total score range: 0-24, higher score=greater severity.
Time Frame: Baseline
Population: SAF population included all participants who signed the informed consent, had exposure to open label study drug and had at least one safety assessment. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Number analyzed (Participants) | 107 | 108
participants
  Little interest in things: Not at All | 59 | 67
  Little interest in things: Several Days | 31 | 25
  Little interest in things: More Than Half the Days | 14 | 9
  Little interest in things: Nearly Every Day | 3 | 7
  Feeling down: Not at All | 84 | 79
  Feeling down: Several Days | 18 | 21
  Feeling down: More Than Half the Days | 5 | 6
  Feeling down: Nearly Every Day | 0 | 2
  Trouble with sleep: Not at All | 57 | 59
  Trouble with sleep: Several Days | 33 | 40
  Trouble with sleep: More Than Half the Days | 14 | 4
  Trouble with sleep: Nearly Every Day | 3 | 5
  Feeling tired: Not at All | 52 | 53
  Feeling tired: Several Days | 43 | 40
  Feeling tired: More Than Half the Days | 12 | 14
  Feeling tired: Nearly Every Day | 0 | 1
  Poor appetite/overeating: Not at All | 75 | 71
  Poor appetite/overeating: Several Days | 24 | 26
  Poor appetite/overeating: More Than Half the Days | 5 | 5
  Poor appetite/overeating: Nearly Every Day | 3 | 6
  Feeling bad about self: Not at All | 92 | 88
  Feeling bad about self: Several Days | 12 | 13
  Feeling bad about self: More Than Half the Days | 2 | 3
  Feeling bad about self: Nearly Every Day | 1 | 4
  Trouble concentrating: Not at All | 79 | 84
  Trouble concentrating: Several Days | 23 | 20
  Trouble concentrating: More Than Half the Days | 2 | 3
  Trouble concentrating: Nearly Every Day | 3 | 1
  Move or speak slow/fidgety: Not at All | 87 | 86
  Move or speak slow/fidgety: Several Days | 18 | 16
  Move or speak slow/fidget: More Than Half the Days | 0 | 3
  Move or speak slow/fidgety: Nearly Every Day | 2 | 3

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin-Pregabalin | Placebo-Pregabalin
Serious Adverse Events (participants affected / at risk) | 4/108 | 3/109
Other Adverse Events (participants affected / at risk) | 35/108 | 50/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin-Pregabalin (N=108) | Placebo-Pregabalin (N=109)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin-Pregabalin (N=108) | Placebo-Pregabalin (N=109)
Oedema peripheral (General disorders) | 2 | 6
Influenza (Infections and infestations) | 5 | 7
Pharyngitis (Infections and infestations) | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 10 | 19
Headache (Nervous system disorders) | 5 | 8
Somnolence (Nervous system disorders) | 9 | 14

LIMITATIONS AND CAVEATS:
The parent double blind trial A0081244 (NCT01049217) was stopped at interim analysis due to lack of efficacy and therefore this open label extension study was also terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.